CLINICAL TRIAL: NCT05486741
Title: Retinal Nerve Fiber Layer Thickness and Macular Thinckness in Myopia, Hyperopia and Emmetropia : An OCT Study
Brief Title: Retinal Nerve Fiber Layer Thickness and Macular Thickness in Myopia, Hyperopia and Emmetropia : An OCT Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mirna Tawab Saied, Doctor, Assiut University
Other Study IDs: OCT study in refractive errors
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: OCT Study RNFL and Macular Thickness
Keywords: OCT study

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Myopes: myopes (≤ -1.0 D)
  Interventions: Other: Optical cehernce tomography
- Hyperopes: hyperopia (≥ +1.0D).
  Interventions: Other: Optical cehernce tomography
- Emmetropes: emmetropes (> -1.0 to <
  * 1.0 D)
  Interventions: Other: Optical cehernce tomography

INTERVENTIONS:
Other: Optical cehernce tomography — OCT macula and disc

SUMMARY:
The purpose of this study is to investigate the variability of RNFL and macular thickness between myopia , hyper metropia and emmetropia

DETAILED DESCRIPTION:
The world health organization (WHO) has estimated that the visual impairment caused by uncorrected refractive errors to be present in 153 million people worldwide (1) the prevalence of myopia ranges from 22.7% to 38.7% in large population study According to the WHO regions the estimated prevalence (EP) of hyperopia is 30.6% with the lowest EP in south east Asia 2.2% and the highest EP in the Americas 14.3% (2-3) During optic nerve development 2.85 million nerve fibers exist but by the third trimester we lose about 35% of these fibers (4) and the perpapillary retinal nerve fiber layer (RNFL) thickness will continue to decrease with advancing age (5). The relationship of the RNFL thickness with the refractive errors has been extensively investigated in adults and in children (6) and there was significant increase in the RNFL thickness in hypermetrope than in emmetrope and myope Understanding the derminants that affect the RNFL reserve helps us in the diagnosis and monitoring of optic nerve diseases. In macular region the thickness measured through optocal coherent tomography OCT shows high variability with value ranging from 190mm (centerpoint) to 389 mm (superior inner/nasal inner macula) (7) for both retinal and macular regions while decreasing in the retinal thickness has been reported with increasing age. Different studies have shown racial differences in RNFL thickness (8) white race (9) and myopia which has high prevelance in East Asian regions (10-12) have been associated with thinner RNFL (11) on the contrary Asian or Hispanic race has been associated with a thicker RNFL

ELIGIBILITY:
Inclusion Criteria:

* All individuals having similar type of refractive status in both eyes and with no known confounding factor affecting retinal intensity or CDVA and willing to participate.

Exclusion Criteria:

* • Eyes with amplyopia

  * Patients having posterior segment pathology or media opacity
  * Patients with history of glaucoma
  * History of retinal laser therapy
  * History of ocualr trauma
  * Any medical disease that prevents patients from positioning on the device

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with errors of refraction devided into 3 groups myopes (≤ -1.0 D) ; emmetropes (> -1.0 to <
  * 1.0 D) and hypermetropia (≥ +1.0D).
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Retinal nerve fiber layer thickness and macular thickness in myopia , hyperopia and emmetropia : An OCT study | Baseline
  investigate the variability of RNFL and macular thickness between myopia , hyper metropia and emmetropia The peripapillary RNFL thickness in central ,perimacular and paramacular regions will be measured using the OCT and compared between three groups of refractive states

REFERENCES:
- [Background] Hussein M, Ibrahim S, Taha A, Magdy R. The impact of error of refraction and retinal nerve fiber layer thickness on cognitive functions in adults with bilateral myopia. Int J Neurosci. 2023 Mar;133(3):290-295. doi: 10.1080/00207454.2021.1910260. Epub 2021 May 17. PMID 33781167
- [Background] Leung CK, Mohamed S, Leung KS, Cheung CY, Chan SL, Cheng DK, Lee AK, Leung GY, Rao SK, Lam DS. Retinal nerve fiber layer measurements in myopia: An optical coherence tomography study. Invest Ophthalmol Vis Sci. 2006 Dec;47(12):5171-6. doi: 10.1167/iovs.06-0545. PMID 17122099
- [Background] Wang Q, Klein BE, Klein R, Moss SE. Refractive status in the Beaver Dam Eye Study. Invest Ophthalmol Vis Sci. 1994 Dec;35(13):4344-7. PMID 8002254